CLINICAL TRIAL: NCT02199899
Title: A Single Increasing Dose Safety, Tolerability and Pharmacodynamics (Citric Acid Challenge) Study After Oral Administration of BIIF 1149 BS (Drinking Solution, Single Doses: 0.1 - 25 mg; in Addition, at 25 mg Also as a 25 mg Tablet) in Healthy Young Male Volunteers (Randomised, Double-blind, Placebo-controlled, Parallel Groups)
Brief Title: Safety, Tolerability and Pharmacodynamics of BIIF 1149 BS in Healthy Young Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1157.2
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIIF 1149 BS - single rising doses (Experimental): BIIF 1149 BS oral drinking solution and a BIIF 1149 BS tablet
  Interventions: Drug: BIIF 1149 BS - single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIF 1149 BS - single rising doses
  Arms: BIIF 1149 BS - single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety and tolerability of BIIF 1149 BS, to determine the pharmacologically active dose (range) by performing a citric acid challenge test and to obtain preliminary pharmacokinetic data

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy males
* Age range from 21 to 50 years
* Within +- 20% of their normal weight (Broca-Index)
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteer is supposed to give his written informed consent prior to admission to the study
* Each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead Electrocardiogram (ECG)
* A citric acid provocation test will be performed to determine the cumulative dose of citric acid which causes at least three coughs. If there will not be at least three coughs after inhalation up to the highest citric acid concentration of 32 % the volunteer will be replaced by a new person
* Haematopoietic, hepatic and renal function test will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (especially respiratory infections, cough)
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>= 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Use of any other drugs which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 40g/day)
* Drug abuse
* Blood donation (>= 100 ml) within the last 4 weeks
* Excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 1999-03; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 4 months

SECONDARY OUTCOMES:
AUC (Area under the concentration-time curve of the analyte in plasma) | up to 120 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 120 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 120 hours after drug administration
Ae (Amount of parent drug excreted into urine) | up to 120 hours after drug administration
MRT (Mean residence time of the analyte in the body) | up to 120 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 120 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 120 hours after drug administration
Ae (amount of analyte excreted into Urine) | up to 120 h after drug administration
CLren (renal clearance) | up to 120 h after drug administration